CLINICAL TRIAL: NCT07241793
Title: A Phase II Clinical Study of Trastuzumab Rezetecan (SHR-A1811) or in Combination With Adebrelimab (SHR-1316) for HER2-Expressing Locally Advanced or Metastatic Urothelial Carcinoma (la/mUC)
Brief Title: Phase II Study of Trastuzumab Rezetecan or in Combination With Adebrelimab in HER2-Expressing Locally Advanced or Metastatic Urothelial Carcinoma (la/mUC)
Acronym: TRAIN-UC-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: The fifth Affiliated Hospital of Guangzhou Medcial University (Other Government); The Second Affiliated Hospital of Kunming Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology (Unknown)
Responsible Party: Principal Investigator, Shi Yanxia, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-281
Record Dates: First submitted 2025-09-24; First posted 2025-11-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Urothelial Carcinoma; Advanced Urothelial Carcinoma; Urothelial Carcinoma Recurrent
Keywords: Urothelial carcinoma; Antibody-Drug Conjugate; immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Study Design:
  Cohort 1: Patients with locally advanced or metastatic UC (la/mUC) who have previously received at least one systemic treatment or experienced relapse/progression within 12 months following the last treatment, or those who are unable to tolerate treatment due to adverse events.
  Cohort 2: Patients with locally advanced or metastatic UC (la/mUC) who have not received prior systemic therapy or who have relapsed/progressed more than 12 months after receiving neoadjuvant/adjuvant therapy, or those who cannot tolerate treatment due to adverse events.
  Cohort 3: Patients with locally advanced or metastatic UC (la/mUC) who have previously been treated with platinum-based chemotherapy (including cisplatin, carboplatin), immune checkpoint inhibitors (such as PD-1, PD-L1 inhibitors), and Disitamab Vedotin .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1:Adebrelimab and Trastuzumab Rezetecan in Patients with Prior Systemic Therapy (Experimental): Patients with locally advanced or metastatic UC (la/mUC) who have previously received at least one systemic treatment or experienced relapse/progression within 12 months following the last treatment, or those unable to tolerate treatment due to adverse events.
  Interventions: Drug: Adebrelimab; Drug: Trastuzumab Rezetecan
- Cohort 2: Adebrelimab and Trastuzumab Rezetecan in Treatment-Naive or Relapsed Patients (Experimental): Patients locally advanced or metastatic UC (la/mUC) who have not received prior systemic therapy or who have relapsed/progressed more than 12 months after receiving neoadjuvant/adjuvant therapy, or those who cannot tolerate treatment due to adverse events.
  Interventions: Drug: Adebrelimab; Drug: Trastuzumab Rezetecan
- Cohort 3: Trastuzumab Rezetecan in Patients with Prior Platinum and Immune Therapy (Experimental): Patients locally advanced or metastatic UC (la/mUC) who have previously been treated with platinum-based chemotherapy (including cisplatin, carboplatin), immune checkpoint inhibitors (such as PD-1, PD-L1 inhibitors), and Disitamab Vedotin .
  Interventions: Drug: Trastuzumab Rezetecan

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab (1200 mg) every 3 weeks (Q3W).
  Arms: Cohort 1:Adebrelimab and Trastuzumab Rezetecan in Patients with Prior Systemic Therapy; Cohort 2: Adebrelimab and Trastuzumab Rezetecan in Treatment-Naive or Relapsed Patients
Drug: Trastuzumab Rezetecan — Trastuzumab Rezetecan (4.8 mg/kg) every 3 weeks (Q3W).

SUMMARY:
This is a multicenter, open-label, Phase II clinical trial to evaluate the efficacy and safety of Trastuzumab Rezetecan (SHR-A1811) or in combination with Adebrelimab (SHR-1316) for HER2-expressing locally advanced or metastatic urothelial carcinoma (la/mUC).

DETAILED DESCRIPTION:
This multicenter Phase II study aims to investigate the clinical efficacy and safety of Trastuzumab Rezetecan (SHR-A1811) or in combination with Adebrelimab (SHR-1316) for HER2-expressing locally advanced or metastatic urothelial carcinoma (la/mUC). The study includes three cohorts based on their prior treatment history and relapse/progression status: Cohort 1 includes patients who have received at least one prior systemic therapy and relapsed/progressed within 12 months; Cohort 2 includes patients who have not received prior systemic therapy or relapsed/progressed more than 12 months after neo-adjuvant/adjuvant treatment; Cohort 3 includes patients who have previously received platinum-based chemotherapy, immunotherapy, or Disitamab Vedotin. The study will provide important data on the combination therapy of Trastuzumab Rezetecan and Adebrelimab, potentially offering a new treatment option for patients with HER2-expressing advanced UC .

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study must meet all of the following criteria:

  1. Age ≥ 18 years;
  2. Histologically or cytologically confirmed HER2-expressing locally advanced unresectable (e.g., T4b, or N2-3) or metastatic urothelial carcinoma (la/mUC), including bladder, ureter, renal pelvis, and urethra. HER2 expression is defined as immunohistochemical (IHC) staining results of 1+ to 3+, and must be confirmed by the pathology department of Sun Yat-sen University Cancer Center according to ASCO/CAP guidelines.
  3. Cohort 1: Patients who have received at least one prior systemic therapy, or relapsed/progressed within 12 months after the last treatment, or who could not tolerate treatment due to adverse events (AEs). Cohort 2: Patients who have not received prior systemic therapy or relapsed/progressed more than 12 months after neoadjuvant/adjuvant therapy, or those who could not tolerate treatment due to AEs. Cohort 3: Patients who have previously received platinum-based chemotherapy (including cisplatin, carboplatin, etc.), immunotherapy (including PD-1, PD-L1 inhibitors), and Disitamab Vedotin ;
  4. At least one measurable target lesion according to RECIST 1.1 criteria;
  5. ECOG performance status ≤ 2;
  6. Adequate bone marrow, renal (calculated creatinine clearance > 30 mL/min using the CG formula), hepatic, and coagulation function;
  7. Expected survival ≥ 3 months;
  8. The patient understands the study procedures and has provided written informed consent to participate in the study;
  9. Female participants of childbearing potential must have a negative urine or serum pregnancy test within 7 days before the first administration of the study drug (Cycle 1, Day 1). If the urine pregnancy test is inconclusive, a blood pregnancy test is required.
  10. Both male and female participants must agree to use highly effective contraception (i.e., methods with a failure rate of less than 1% per year) and continue contraception until at least 180 days after the end of study treatment.

Exclusion Criteria:

1. Locally advanced patients who are candidates for curative local treatment;
2. Clinical history of cardiovascular, liver, respiratory, renal, hematological, endocrine, or neurological/psychiatric diseases;
3. Known or untreated spinal cord compression or active central nervous system metastases, except for those who have been treated and stable for at least 1 month and have discontinued corticosteroids for > 2 weeks;
4. Known severe allergic reactions to the study drug's active ingredients and/or excipients, or allergy to humanized monoclonal antibody products (e.g., trastuzumab, pertuzumab);
5. Received antitumor monoclonal antibody treatment within 4 weeks before the study start, or received other antitumor therapy without recovery from adverse events;
6. Participated in any investigational drug treatment within 4 weeks before the study started;
7. Known or suspected interstitial lung disease, or moderate to severe pulmonary diseases that might interfere with the evaluation of drug-related pulmonary toxicity, including but not limited to idiopathic pulmonary fibrosis, organizing pneumonia, bronchitis obliterans, pulmonary embolism, severe asthma, COPD, restrictive pulmonary diseases, or any autoimmune, connective tissue or inflammatory lung diseases, such as rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc., or a history of total lung resection;
8. Known hereditary or acquired bleeding disorders (e.g., hemophilia, coagulopathy);
9. Received spinal cord radiation or has not recovered from radiation-related adverse events within 4 weeks before study start;
10. Diagnosed with immunodeficiency or received systemic corticosteroid treatment or any other immunosuppressive therapy within 7 days before the first study drug administration. Physiological doses of corticosteroids (≤10 mg/day of prednisone or equivalent) are allowed;
11. Active autoimmune diseases requiring systemic treatment within the past 2 years (e.g., requiring disease-modifying drugs, corticosteroids, or immunosuppressants). Replacement therapies (e.g., thyroid hormones, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatments. A history of non-infectious pneumonia requiring corticosteroid treatment or current interstitial lung disease within 1 year before the first dose is excluded;
12. History of organ or hematopoietic stem cell transplantation;
13. Known HIV infection (HIV 1/2 positive);
14. Untreated active hepatitis B (HBV). Note: Hepatitis B carriers with an HBV viral load < 1000 copies/mL (200 IU/mL) before the first dose are eligible, but should receive antiviral therapy during chemotherapy to prevent reactivation.

    For anti-HBc (+), HBsAg (-), anti-HBs (-), and undetectable HBV viral load subjects, preventive antiviral therapy is not required, but close monitoring is necessary.
15. Active hepatitis C (HCV) infection (HCV antibody positive and HCV RNA level above detection threshold;
16. Received live vaccines within 30 days before the first dose of the study drug. Note: Inactivated flu vaccines are allowed within 30 days before the first dose, but live attenuated flu vaccines are not permitted.
17. History of other malignancies within the past 3 years, except for cured non-melanoma skin cancer, cervical carcinoma in situ, or low-risk prostate cancer (T2N0M0, Gleason score <7, or undetectable PSA);
18. Any condition or disease history that may interfere with the study results or hinder the participant's full participation, including abnormal laboratory values, or situations deemed inappropriate by the investigator;
19. Breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Within approximately 36 months
  Objective Response Rate (ORR) is defined as the proportion of participants achieving a complete response (CR) or partial response (PR) as determined by RECIST v1.1 criteria, based on radiologic assessment. Responses will be confirmed by at least one subsequent imaging assessment.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Within approximately 36 months
  Progression-Free Survival (PFS) is defined as the time from the first dose of study treatment to the first documented disease progression, as determined by RECIST v1.1, or death from any cause, whichever occurs first. Disease progression will be assessed by independent radiologic review. Patients without documented progression or death at the time of analysis will be censored at their last tumor assessment date.
Overall Survival (OS) | Within approximately 36 months
  Overall Survival (OS) is defined as the time from the first dose of study treatment to death from any cause. Participants still alive at the time of analysis will be censored at the date of their last follow-up.
Disease Control Rate (DCR) | Within approximately 36 months
  Disease Control Rate (DCR) is defined as the proportion of participants achieving a complete response (CR), partial response (PR), or stable disease (SD) for at least 6 weeks after treatment initiation, based on RECIST v1.1 criteria.
Time to Response (TTR) | Within approximately 36 months
  Time to Response (TTR) is defined as the time from the first dose of study treatment to the first occurrence of a confirmed objective response (CR or PR) as determined by RECIST v1.1 criteria.
Duration of Response (DOR) | Within approximately 36 months
  Duration of Response (DOR) is defined as the time from the first documented objective response (CR or PR) to disease progression or death, whichever occurs first, based on RECIST v1.1 criteria.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Within approximately 36 months
  The number of participants who experience treatment-related adverse events (AEs) will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. AEs will be graded on a scale from Grade 1 (mild) to Grade 5 (death related to AE). The severity, frequency, and type of AEs will be recorded and summarized. The results will be presented as the total number and percentage of participants experiencing any treatment-related AE, as well as a breakdown by AE grade and type. Treatment-related AEs will be determined by the investigator's clinical judgment based on available data.
Health-Related Quality of Life (HRQoL) as Assessed by the EORTC QLQ-C30 Questionnaires | Within approximately 36 months
  The EORTC QLQ-C30 will assess global health status, physical and emotional functioning, and cancer-related symptoms such as fatigue, pain, nausea, and appetite loss. The tool also evaluates functional scales across physical, role, emotional, cognitive, and social domains. The QLQ-C30 is a widely validated tool for cancer patients' HRQoL assessment.
  Scores for each domain range from 0 to 100. Each functional domain score (physical, role, emotional, cognitive, and social) is calculated by averaging the responses for the items within that domain. Symptom domain scores (e.g., fatigue, pain) are also calculated by averaging their respective items. A higher score for symptom domains indicates worse quality of life, while a higher score for functional domains indicates better quality of life.
Health-Related Quality of Life (HRQoL) as Assessed by the EQ-5D | Within approximately 36 months
  Health-related quality of life will be assessed using the EQ-5D, which is a standardized tool for measuring general health status. The EQ-5D assesses five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 3-level scale: 1. No problems ；2. Some problems；3. Extreme problems.
  The EQ-5D index score is calculated based on the responses for each dimension. A higher score indicates better health status. Additionally, the Visual Analog Scale (VAS) will be used, where participants rate their overall health on a scale from 0 (worst imaginable health) to 100 (best imaginable health).

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Shi, Doctor, Principal Investigator — Sun Yat-sen University
Locations (5):
- China (5):
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun yat-sen university cancer center, Guangzhou, Guangdong
  - The fifth Affiliated Hospital of Guangzhou Medcial University, Guangzhou, Guangdong
  - Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical and privacy concerns.